CLINICAL TRIAL: NCT03920215
Title: Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease (The ONSET Study)-Long Term Safety Follow-up
Brief Title: Evaluation of the Long Term Follow up of the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPP-002-01EXT
Record Dates: First submitted 2019-04-09; First posted 2019-04-18 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2021-09

CONDITIONS: Long Term Follow up Dry Eye Disease
MeSH Terms: interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OC-01 Low Dose, 0.12 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 0.12 mg/mL
  Interventions: Drug: OC-01 Low Dose, 0.12 mg/mL
- OC-01 Mid Dose, 0.6 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 0.60 mg/mL
  Interventions: Drug: OC-01 Mid Dose, 0.6 mg/mL
- OC-01 High Dose, 1.2 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 1.2 mg/mL
  Interventions: Drug: OC-01 High Dose, 1.2 mg/mL
- Placebo (vehicle) nasal spray (Placebo Comparator): Placebo (vehicle) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 Low Dose, 0.12 mg/mL — OC-01 (varenicline) nasal spray
  Other Names: OC-01 (varenicline) nasal spray, 0.12 mg/ml
  Arms: OC-01 Low Dose, 0.12 mg/mL
Drug: OC-01 Mid Dose, 0.6 mg/mL — OC-01 (varenicline) nasal spray
  Arms: OC-01 Mid Dose, 0.6 mg/mL
Drug: OC-01 High Dose, 1.2 mg/mL — OC-01 (varenicline) nasal spray
  Other Names: OC-01 Mid Dose, 1.2 mg/mL
  Arms: OC-01 High Dose, 1.2 mg/mL
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
The objective of this safety long-term follow-up study was to evaluate the safety of OC-01 Nasal Spray at 6 months and 12 months post treatment in the OPP-002 study (NCT03636061).

DETAILED DESCRIPTION:
Study OPP-002-01 was a long-term follow-up study of those subjects who had previously participated in the OPP-002 study (NCT03636061). The OPP-002 study is a Phase 2, multicenter, randomized, double-masked, placebo-controlled study designed to evaluate the safety and efficacy of OC-01 nasal spray in adult participants with dry eye disease.

The first scheduled visit occurs 6 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study. The second scheduled visit occurs 12 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study.

ELIGIBILITY:
Inclusion Criteria:

1. Have been enrolled in the OPP-002 study
2. Have received at least one dose of the study drug/placebo in OPP-002 study
3. Completed the OPP-002 study to Visit 5
4. Have provided verbal and written informed consent

Exclusion Criteria:

1. Have discontinued prior to Visit 5 in the OPP-002 study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Newport Beach, Newport Beach, California
  - Indianapolis, Indianapolis, Indiana
  - Andover, Andover, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OC-01 Mid Dose, 0.6 mg/mL: OC-01 (varenicline) nasal spray, 0.62 mg/mL
  OC-01 Mid Dose, 0.6 mg/mL: OC-01 (varenicline) nasal spray
Period: Overall Study
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Started | 26 | 29 | 23 | 23
Completed | 25 | 27 | 23 | 22
Not Completed | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects in the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray | Total
Number analyzed (Participants) | 26 | 29 | 23 | 23 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9.45) | 68.9 (9.25) | 69.8 (6.64) | 63.3 (11.38) | 67.4 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 19 | 16 | 74
  Male | 7 | 9 | 4 | 7 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 23 | 23 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Left Nostril/Abnormal at 6 Months as Assessed by Intranasal Examinations
Description: Number of Participants with the Left Nostril/Abnormal at 6 months as assessed by Intranasal Examinations
Time Frame: 6 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study (Visit 1 OPP-002 and 6 months)
Population: Subjects in the ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 26 | 29 | 23 | 23
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With the Right Nostril/Abnormal at 6 Months as Assessed by Intranasal Examinations
Description: Number of Participants with the Right Nostril/Abnormal at 6 months as assessed by Intranasal Examinations
Time Frame: 6 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study (Visit 1 OPP-002 and 6 months)
Population: Subjects in the ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 26 | 29 | 23 | 23
Participants | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With the Left Nostril/Abnormal at 12 Months as Assessed by Intranasal Examinations
Description: Number of Participants with the Left Nostril/Abnormal at 12 months as assessed by Intranasal Examinations
Time Frame: 12 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study (Visit 1 OPP-002 and 12 months)
Population: Subjects in the ITT population (subjects with non-missing data).
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 25 | 27 | 23 | 22
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With the Right Nostril/Abnormal at 12 Months as Assessed by Intranasal Examinations
Description: Number of Participants with the Right Nostril/Abnormal at 12 months as assessed by Intranasal Examinations
Time Frame: 12 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study (Visit 1 OPP-002 and 12 months)
Population: Subjects in the ITT population (subjects with non-missing data)
Measure: Count of Participants; unit: Participants
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 25 | 27 | 23 | 22
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 months after the first treatment of OC-01 nasal spray/placebo in the OPP-002 study.
Arm/Group | OC-01 Low Dose, 0.12 mg/mL | OC-01 Mid Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/29 | 0/23 | 1/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/29 | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 3/26 | 5/29 | 5/23 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 Low Dose, 0.12 mg/mL (N=26) | OC-01 Mid Dose, 0.6 mg/mL (N=29) | OC-01 High Dose, 1.2 mg/mL (N=23) | Placebo (Vehicle) Nasal Spray (N=23)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 Low Dose, 0.12 mg/mL (N=26) | OC-01 Mid Dose, 0.6 mg/mL (N=29) | OC-01 High Dose, 1.2 mg/mL (N=23) | Placebo (Vehicle) Nasal Spray (N=23)
Conjunctival oedema (Eye disorders) | 0 | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Instillation site pruritis (General disorders) | 0 | 1 | 0 | 0
Device (IOL) dislocation (Product Issues) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT03920215/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT03920215/SAP_001.pdf